CLINICAL TRIAL: NCT03518060
Title: Durability of Antiretroviral Suppression and the Real World Clinical Profile of the Novel 2-Drug Regimen Juluca, a Onepill-Regimen Consisting of Dolutegravir and Rilpivirine, in Routine Clinical Care in Germany
Brief Title: Dolutegravir/Rilpivirine, Antiretroviral Efficacy Study Using Real-world Data in Subjects With Human Immunodeficiency Virus (HIV)-1
Acronym: JUNGLE
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: MUC Research GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 208982
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: 2 drug regimen; Juluca; Rilpivirine; Dolutegravir; Antiretroviral; One pill regimen
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir, rilpivirine drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who received JULUCA: Virologically suppressed HIV positive participants, on a stable antiretroviral regimen, who switched to the 2-Drug Regimen JULUCA (Dolutegravir [DTG] / Rilpivirine [RPV]) were included in the study. Participants were followed-up for approximately 3 years during routine clinical practice.
  Interventions: Drug: JULUCA

INTERVENTIONS:
Drug: JULUCA — JULUCA is a combination of dolutegravir (INSTI) and rilpivirine (NNRTI).

SUMMARY:
This was a prospective, non-interventional, single-arm, multi-center study aimed at gathering real-world data on JULUCA use in routine clinical care in Germany, to supplement clinical trial data to further improve/optimize care in HIV positive participants in Germany. Approximately 250 virologically suppressed HIV positive participants on stable antiretroviral therapy (ART) were included in the study at the discretion of treating physician. Eligible participants were followed up for approximately 3 years and data was collected during routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Greated than or equal to (>=)18 years of age.
* Documented HIV-1 infection.
* Virologically suppressed (HIV-1 ribonucleic acid [RNA] less than [<] 50 copies [c]/mL for at least 6 months)
* Prescription for JULUCA was issued independently from entering this study.
* Ability to understand informed consent form and other relevant study documents

Exclusion Criteria:

* Any contraindication according to JULUCA SmPC.
* Documented viral load greater than (>) 50 c/mL at any time point within 6 months prior to inclusion into this study.
* History of treatment failure.
* Known or suspected substitutions associated with resistance to any non-nucleoside reverse-transcriptase inhibitors (NNRTI) or integrase strand transfer inhibitor (INSTI).
* Any ART for the treatment of HIV-1 in addition to JULUCA.
* Hepatitis B virus (HBV)-co-infection.
* Current participation in the ongoing non-interventional study TRIUMPH (study number: 202033) or any interventional clinical trial irrespective of indication.
* Previous participation in clinical trials involving JULUCA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred treatment experienced and virologically suppressed HIV positive participants were included in this study. The participants were included at the discretion of the treating physician based on the local summary of product characteristics (SmPC) of JULUCA.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (12):
- Germany (12):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bochum
  - GSK Investigational Site, Chemnitz
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
  - GSK Investigational Site, Münster
  - GSK Investigational Site, Osnabrück
  - GSK Investigational Site, Tübingen
  - GSK Investigational Site, Weimar

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 209 participants were enrolled in the full analysis set (FAS) from which 9 participants were excluded due to not meeting the eligibility criteria. Therefore, 200 participants formed the modified FAS (mFAS).
Period: Overall Study
Arm/Group | Participants Who Received JULUCA
Started | 200
Completed | 124
Not Completed | 76
Not completed — Death | 1
Not completed — Poor adherence | 1
Not completed — Withdrawal of informed consent | 2
Not completed — Interaction with comedication or comorbidities | 4
Not completed — Physician Decision | 7
Not completed — Adverse drug reactions | 23
Not completed — Withdrawal by Subject | 25
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 49.0 [40.0 to 57.0]
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 104
  >= 50 years | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 181
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Suppression at Year 3
Description: Virologic suppression (VS) was defined as HIV-RNA less than (<) 50 copies (c)/mL for at least 6 months or, if between 50-200 c/mL with a subsequent next available measurement (within 120 days) <50 c/mL at Year 3 follow-up. Any subsequent measurement was accepted as a consecutive measurement as long as measured no later than 120 days after the initial measurement. If no subsequent HIV-RNA measurement was performed within 120 days, this was scored as a confirmed HIV-RNA greater than or equal to (>=)200 c/mL.
Time Frame: At Year 3
Population: The analysis was performed on the modified Full Analysis Set (mFAS) which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  HIV-RNA <50 c/mL | 119
  HIV-RNA 50-200 c/mL and subsequent measurement <50 c/mL | 2
  HIV-RNA 50-200 copies/mL & subsequent measurement >=50 c/mL | 1
  HIV-RNA 50-200 c/mL & missing subsequent measurement | 1
  Discontinuation due to intolerability & LOCF HIV-RNA <50 c/mL | 23
  Discontinuation due to death & LOCF HIV-RNA <50 c/mL | 1
  Discontinuation due to other reasons & LOCF HIV-RNA <50 c/mL | 35
  Discontinuation due to other reasons & LOCF HIV-RNA >=50 c/mL | 4
  Lost to follow-up & LOCF HIV-RNA <50 c/mL | 13
  On drug, but no HIV-RNA in window & LOCF HIV-RNA <50 c/mL | 1

2. Secondary Outcome: Number of Participants With Sustained Virologic Suppression at Year 1 and Year 2
Description: VS was defined as HIV-RNA <50 c/mL for at least 6 months or, if between 50-200 c/mL with a subsequent next available measurement (within 120 days) <50 c/mL. Any subsequent measurement was accepted as a consecutive measurement as long as measured no later than 120 days after the initial measurement. If no subsequent HIV-RNA measurement was performed within 120 days, this was scored as a confirmed HIV-RNA >=200 c/mL.
Time Frame: At Year 1 and Year 2
Population: The analysis was performed on the mFAS which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  HIV-RNA <50 c/mL - at Year 1 | 164
  HIV-RNA 50-200 c/mL and subsequent measurement <50 c/mL - at Year 1 | 2
  HIV-RNA 50-200 c/mL & subsequent measurement >=50 copies/mL - at Year 1 | 0
  HIV-RNA 50-200 c/mL & missing subsequent measurement - at Year 1 | 1
  HIV-RNA >=200 copies/mL - at Year 1 | 0
  Discontinuation due to intolerability & LOCF HIV-RNA <50 c/mL - at Year 1 | 19
  Discontinuation due to death & LOCF HIV-RNA <50 c/mL - at Year 1 | 1
  Discontinuation due to other reasons & LOCF HIV-RNA <50 c/mL - at Year 1 | 9
  Discontinuation due to other reasons & LOCF HIV-RNA >=50 c/mL - at Year 1 | 0
  Lost to follow-up & LOCF HIV-RNA <50 c/mL - at Year 1 | 3
  On drug, but no HIV-RNA in window & LOCF HIV-RNA <50 c/mL - at Year 1 | 1
  HIV-RNA <50 c/mL - at Year 2 | 143
  HIV-RNA 50-200 c/mL and subsequent measurement <50 c/mL - at Year 2 | 3
  HIV-RNA 50-200 c/mL & subsequent measurement >=50 copies/mL - at Year 2 | 0
  HIV-RNA 50-200 c/mL & missing subsequent measurement - at Year 2 | 0
  HIV-RNA >=200 c/mL - at Year 2 | 1
  Discontinuation due to intolerability & LOCF HIV-RNA <50 c/mL - at Year 2 | 22
  Discontinuation due to death & LOCF HIV-RNA <50 c/mL - at Year 2 | 1
  Discontinuation due to other reasons & LOCF HIV-RNA <50 c/mL - at Year 2 | 17
  Discontinuation due to other reasons & LOCF HIV-RNA >=50 c/mL - at Year 2 | 3
  Lost to follow-up & LOCF HIV-RNA <50 c/mL - at Year 2 | 8
  On drug, but no HIV-RNA in window & LOCF HIV-RNA <50 c/mL - at Year 2 | 2

3. Secondary Outcome: Number of Participants With Low Level Viremia
Description: Low level viremia was defined as a VL greater than (>) 50 to <200 c/mL.
Time Frame: At Year 1, Year 2 and Year 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  HIV-RNA 50-200 c/mL and subsequent measurement >=50 c/mL - at Year 1 | 0
  mHIV-RNA 50-200 c/mL and subsequent measurement >=50 c/mL - at Year 2 | 0
  HIV-RNA 50-200 c/mL and subsequent measurement >=50 c/mL - at Year 3 | 1

4. Secondary Outcome: Number of Participants With Virologic Rebound
Description: Virologic rebound was defined as two consecutive VL measurements of >=200 c/mL.
Time Frame: At Year 1, Year 2 and Year 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  HIV-RNA >=200 c/mL - at Year 1 | 0
  HIV-RNA >=200 c/mL - at Year 2 | 1
  HIV-RNA >=200 c/mL - at Year 3 | 0

5. Secondary Outcome: Number of Participants With Treatment Switch
Description: The treatment switch could have been due to virologic failure (VF) or due to intolerability and last observation carried forward (LOCF) as determined at the discretion of the physician.
Time Frame: At Year 1, Year 2 and Year 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  Discontinuation due to intolerability and LOCF HIV-RNA <50 c/mL - at Year 1 | 19
  Discontinuation due to intolerability and LOCF HIV-RNA <50 c/mL - at Year 2 | 22
  Discontinuation due to intolerability and LOCF HIV-RNA <50 c/mL - at Year 3 | 23

6. Secondary Outcome: Number of Monitoring Measures During the 3-year Follow-up
Description: The HIV monitoring measures included were defined as HIV-RNA measurements, normalized to participant years.
Time Frame: Up to Year 3
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Measurements per year
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Measurements per year | 4 [3.6 to 4.4]

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal investigational product, whether or not related to the medicinal investigational product.
  A SAEs was defined as any adverse event meeting the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a congenital anomaly in the off-spring of a participant, was medically significant or could have required intervention to prevent the previously stated outcomes.
Time Frame: Up to Year 3
Population: The analysis was performed on the safety analysis set (SAS) which included all participants who received at least one dose of DTG+RPV.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants | 52

8. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: An ADR was defined as a noxious and unintended response to a medicinal investigational product related to any dose where at least a reasonable possibility (i.e. the relationship) cannot be ruled out.
Time Frame: Up to Year 3
Population: The analysis was performed on the SAS which included all participants who received at least one dose of DTG+RPV.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants | 41

9. Secondary Outcome: Number of Participants With Adherence to Therapy
Description: Adherence to therapy refers to the missed monthly doses. At each follow-up visit, participants were asked to give an estimation of their level of adherence to their antiretroviral therapy (ART).
Time Frame: At Year 1, Year 2 and Year 3
Population: The analysis was performed on the mFAS which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations. This analysis was performed only on the participants from the mFAS who completed the self-assessment questionnaire of adherence.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 174
Participants
  Year 1 | 111
  Year 2: number analyzed (Participants) | 148
  Year 2 | 109
  Year 3: number analyzed (Participants) | 124
  Year 3 | 87

10. Secondary Outcome: Change From Baseline (BL) in Lipid Laboratory Values
Description: To assess the impact on the lipid metabolism, changes in the following parameters were analyzed: total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides.
Time Frame: At Year 1, Year 2 and Year 3
Population: The analysis was performed on the mFAS which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations. This analysis was performed only on the participants from the mFAS who had laboratory parameters data at baseline and at years 1, 2 or 3.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 154
mg/dL
  Change in total cholesterol from BL - at Year 1 | -2.5 [-23 to 19]
  Change in LDL cholesterol from BL - at Year 1: number analyzed (Participants) | 139
  Change in LDL cholesterol from BL - at Year 1 | 1 [-13.5 to 18]
  Change in HDL cholesterol from BL - at Year 1: number analyzed (Participants) | 133
  Change in HDL cholesterol from BL - at Year 1 | -0.8 [-5.8 to 3.1]
  Change in triglycerides from BL - at Year 1: number analyzed (Participants) | 142
  Change in triglycerides from BL - at Year 1 | -1.4 [-56 to 34]
  Change in total cholesterol from BL - at Year 2: number analyzed (Participants) | 131
  Change in total cholesterol from BL - at Year 2 | -3 [-24 to 19]
  Change in LDL cholesterol from BL - at Year 2: number analyzed (Participants) | 121
  Change in LDL cholesterol from BL - at Year 2 | 7 [-17 to 21]
  Change in HDL cholesterol from BL - at Year 2: number analyzed (Participants) | 113
  Change in HDL cholesterol from BL - at Year 2 | -1.4 [-6 to 4]
  Change in triglycerides from BL - at Year 2: number analyzed (Participants) | 124
  Change in triglycerides from BL - at Year 2 | 3.5 [-38.5 to 49.3]
  Change in total cholesterol from BL - at Year 3: number analyzed (Participants) | 107
  Change in total cholesterol from BL - at Year 3 | -5 [-27 to 18]
  Change in LDL cholesterol from BL - at Year 3: number analyzed (Participants) | 99
  Change in LDL cholesterol from BL - at Year 3 | -1.9 [-21 to 20]
  Change in HDL cholesterol from BL - at Year 3: number analyzed (Participants) | 94
  Change in HDL cholesterol from BL - at Year 3 | -2 [-5.8 to 3.9]
  Change in triglycerides from BL - at Year 3: number analyzed (Participants) | 100
  Change in triglycerides from BL - at Year 3 | -1 [-46.5 to 47]

11. Secondary Outcome: Change in Treatment Satisfaction
Description: The change in HIV treatment satisfaction was assessed with the help of the HIV Treatment Satisfaction questionnaire (HIVTSQs), which is a 10-item-self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility, etc. HIV TSQs total score: unweighted sum of 10 items of the HIV TSQs (range: 0-60; with higher scores indicating greater treatment satisfaction).
Time Frame: At Year 1, Year 2 and Year 3
Population: The analysis was performed on the mFAS which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations. This analysis was performed only on the participants from the mFAS who completed the HIV TSQs.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 112
Score on a scale
  Year 1 | 1 [0 to 5.5]
  Year 2: number analyzed (Participants) | 82
  Year 2 | 2.5 [0 to 7]
  Year 3: number analyzed (Participants) | 68
  Year 3 | 3 [0 to 9]

12. Secondary Outcome: Change in Symptom Distress
Description: The change in HIV symptom distress was assessed with the help of the HIV Symptom Distress Module (SDM); which is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. SDM total score: unweighted sum of the 20 items (using a 5-point scale, ranging from 0-4), ranging from 0 to 80. Higher scores indicate higher degrees of symptom distress.
Time Frame: At Year 1, Year 2 and Year 3
Population: The analysis was performed on the mFAS which included all eligible participants who did not have any violation of inclusion or exclusion criteria which also included screening failures and major protocol deviations. This analysis was performed only on the participants from the mFAS who completed the HIV SDM.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 109
Score on a scale
  Year 1 | 0 [-6 to 4]
  Year 2: number analyzed (Participants) | 86
  Year 2 | -1 [-8 to 2]
  Year 3: number analyzed (Participants) | 68
  Year 3 | -1.5 [-6 to 3.5]

13. Secondary Outcome: Number of Participants by Reasons for Therapy Switch to JULUCA
Description: The primary and secondary reasons for therapy switch were presented.
Time Frame: At Baseline (Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received JULUCA
Number analyzed (Participants) | 200
Participants
  Side effects of previous ART | 53
  Potential/real interactions | 8
  Reduction in number of drugs | 41
  Non-nucleoside reverse transcriptase inhibitor (NRTI) - free regime | 9
  Pill size | 1
  Simplification to a single-tablet regimen | 45
  Patient's preference | 24
  Other | 19

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs) and All-Cause Mortality were collected from Day 1 up to maximum Year 3.
Arm/Group | Participants Who Received JULUCA
All-Cause Mortality (participants affected / at risk) | 1/200
Serious Adverse Events (participants affected / at risk) | 52/200
Other Adverse Events (participants affected / at risk) | 41/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received JULUCA (N=200)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myopericarditis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Drug ineffective (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Acute hepatitis B (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Angiogram (Investigations) | 1 (1)
Continuous glucose monitoring (Investigations) | 1 (1)
Nitrite urine (Investigations) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal cavity drainage (Surgical and medical procedures) | 1 (1)
Cardioversion (Surgical and medical procedures) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Mitral valve repair (Surgical and medical procedures) | 2 (2)
Shoulder operation (Surgical and medical procedures) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received JULUCA (N=200)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Sleep disorder (Psychiatric disorders) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03518060/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03518060/SAP_001.pdf